CLINICAL TRIAL: NCT05109299
Title: Antibacterial Effect of Miswak Toothpaste Compared to Fluoride Toothpaste in High Caries Risk Patients: Randomized Clinical Trial
Brief Title: Antibacterial Effect of Miswak Toothpaste Compared to Fluoride Toothpaste
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Osama Shaalan, Lecturer, Conservative Dentistry Department, Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: miswak
Record Dates: First submitted 2021-10-15; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Caries
Keywords: Antibacterial, streptococcus mutans, miswak, fluoride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Miswak toothpaste (Experimental): Dabur meswak herpal toothpaste
  Interventions: Other: Miswak toothpaste
- Fluoride toothpaste (Active Comparator): Signal fluoride toothpaste, containing 1450 ppm of fluoride
  Interventions: Other: Fluoride toothpaste

INTERVENTIONS:
Other: Miswak toothpaste — Dabur Meswak is scientifically formulated herbal toothpaste with pure extract of the Miswak plant 'Salvadore Persica'
  Other Names: Dabur meswak
  Arms: Miswak toothpaste
Other: Fluoride toothpaste — 1450 ppm fluoride toothpaste
  Other Names: Signal toothpaste
  Arms: Fluoride toothpaste

SUMMARY:
Meswak is scientifically formulated herbal toothpaste with pure extract of the Miswak plant 'Salvadore Persica', the famous 'Toothbrush Tree' used for centuries. The astringent and anti-bacterial properties of Meswak helps reduce tooth decay , fight plaque and prevent gum diseases. Miswak Herb is a rare, potent, priceless, wonder herb that delivers incredible Dental Care benefits.

DETAILED DESCRIPTION:
This study is a randomized clinical trial, with parallel study design, 1:1 allocation ratio and superiority framework. The aim of the current trial is to evaluate antibacterial effect miswak toothpaste compared to fluoride toothpaste in high caries risk patients.

ELIGIBILITY:
Inclusion Criteria:

* High caries risk patients.
* At least one carious tooth according to CAT caries risk assessment model.
* Patient compliance

Exclusion Criteria:

* Participant in another trial.
* Using another antimicrobial agents since one month of sampling.
* Systemic diseases or concomitant medication affecting salivary flow.
* Parafunctional habits.
* Pregnancy.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
streptococcus mutans count | 3 months
  Counting streptococcus mutans, Measurement: Mitis-Salivarius agar plate, Unit: CFUs/mL

CONTACTS AND LOCATIONS:
Overall Officials: Omar O Shaalan, PhD, Principal Investigator — Lecturer, Conservative Dentistry Department, Faculty of Dentistry, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, El Manial, Egypt

IPD SHARING:
Plan to Share IPD: No